CLINICAL TRIAL: NCT04721678
Title: INDIGO - Internet-administered Interpersonal Psychotherapy for Depressive Symptoms
Brief Title: Internet-administered Interpersonal Psychotherapy for Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INDIGO
Record Dates: First submitted 2021-01-08; First posted 2021-01-25 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder
Keywords: Interpersonal Psychotherapy; Major Depressive Disorder; Internet Intervention; Internet-based psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal psychotherapy (IPT) (Experimental): 10 weeks of internet-administered interpersonal psychotherapy with therapist support.
  Interventions: Behavioral: Interpersonal psychotherapy
- Wait-list control group (No Intervention): The participants in the control group will receive access to the treatment after the post-treatment assessment has been conducted.

INTERVENTIONS:
Behavioral: Interpersonal psychotherapy — Internet-based interpersonal psychotherapy aimed at reducing symptoms of depression. The content of the intervention is divided into three parts: the assessment phase (the first four weeks), the focus phase (the following five weeks), and the end phase (the last week).
  Arms: Interpersonal psychotherapy (IPT)

SUMMARY:
The aim of the study is to test the efficacy of a treatment for depression based on interpersonal psychotherapy (IPT). The treatment will be accessed via an internet platform built for this study. A therapist will provide support weekly, as well as on-demand when needed. The treatment lasts for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Major depressive disorder (as indicated by the MINI 7.0 Neuropsychiatric interview) and/or depressive symptoms equal to or more severe than mild depression on the MADRS-S (equal to or above 13 points) and/or BDI (equal to or above 14 points).
* Age of at least 18 years old.
* Adequate ability to speak, write, and read Swedish.
* Internet access for the duration of the study.

Exclusion Criteria:

* Ongoing substance abuse.
* Suicidal plans.
* A diagnosed personality syndrome (as diagnosed before the study by a licensed psychiatric healthcare professional).
* Other ongoing psychological treatment.
* Other severe psychiatric comorbidity that requires specialized care (e.g. anorexia nervosa, psychosis).
* Recent changes in psychotropic medication or planned changes during the initial treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change on Montgomery Åsberg Depression Rating Scale (MADRS-S) | Before the treatment, during week 1 to 10 of the treatment, after 11 weeks. Follow-up one year after the start of the treatment.
  Depression inventory, consists of 9 items measuring symptoms of major depressive disorder. Each item are scored between 0 and 6 points, resulting in a total sum between 0 and 54. Cut-offs are: 0-12 No substantial depressive symptoms, 13-19 mild depressive symptoms, 20-34 moderate depressive symptoms, 35-54 severe depressive symptoms.

SECONDARY OUTCOMES:
Change on Beck Depression Inventory-II (BDI-II) | Before treatment and after 11 weeks, follow-up one year after the start of the treatment.
  Depression inventory consisting of 21 items measuring symptoms of depressions along with behavioural and cognitive manifestations of these symptoms. Sum scores range between 0 and 63 points. Cut-offs: 0-13 minimal depressive symptoms, 14-19 mild depressive symptoms, 20-28 moderate depressive symptoms, 30-63 severe depressive symptoms.
Change on Brunnsviken Brief Quality of Life Inventory (BBQ) | Before treatment and after 11 weeks, follow-up one year after the start of the treatment.
  Measure of subjective quality of life. Sum scores can range between 0 and 96. Higher scores indicate a higher quality of life.
Change on Generalized Anxiety Disorder 7-Item Scale (GAD-7) | Before treatment and after 11 weeks, follow-up one year after the start of the treatment.
  Seven item measure of generalized anxiety disorder. Sum score range from 0 to 21, with higher scores indicating more generalized anxiety. Cut-offs for interpretation: 0-5 minimal anxiety, 6-9 mild anxiety, 10-14 moderate anxiety, and 15-21 severe anxiety.
Change on Reflective Functioning Questionnaire-8 item version (RFQ-8) | Before treatment, after 11 weeks, following one year after the start of the treatment.
  Instrument measuring reflective functioning related to mentalization ability. Eight items where the respondent answers on a Likert scale. The scoring is calculated based on two scales, uncertainty and certainty. All eight items are scored twice, once for each scale. The Likert options for the scoring of the first scale is scored 0 0 0 0 1 2 3. The same items are then summed again with the scoring 3 2 1 0 0 0 0. All items are the summed up to give a measure of mentalization certainty and uncertainty.

OTHER OUTCOMES:
Change on The Medical Outcome Social Support Survey, 12-item short form (MOS-SSS) | Before the treatment, during week 1 to 10 of the treatment, after 11 weeks.
  Mediational measure of perceived social support. Consists of six items summed up to a score between 12 and 60. Higher scores indicate more perceived social support.
Score on Interpersonal Psychotherapy Outcome Scale (IPOS) | Measured 11 weeks after the start of the intervention.
  Questionnaire asking the participant to identify the focus of the treatment and the perceived change in each focus area. Change is measured on a five-point Likert scale ranging from worsened significantly to improved greatly.
Score on Credibility and Expectancy Questionnaire (CEQ) | Measured during week 3 of the intervention.
  Measure of the credible the participant perceive the intervention to be as well as how beneficial they expect it to be. Consists of six items, with four of them being answered on a nine-point Likert scale and two responses given on a ten-point Likert scale. Scores can range between 4 and 56, with higher scores indicating greater credibility and expectancy of positive change during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kall A, Back M, Fahlroth O, Ekeflod E, Lundberg A, Viberg N, Andersson G. Internet-based therapist-supported interpersonal psychotherapy for depression: A randomized controlled trial. J Affect Disord. 2025 Jan 15;369:188-194. doi: 10.1016/j.jad.2024.09.171. Epub 2024 Sep 27. PMID 39343313